CLINICAL TRIAL: NCT05402449
Title: To Evaluate the Clinical Efficacy of Probiotic in Patients With NAFLD
Brief Title: To Evaluate the Beneficial Effect of Probiotics on NAFLD Patients and the Role of Gut Microbiota Modulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GenMont Biotech Incorporation (Industry)
Collaborators: Fu Jen Catholic University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NAFLD2022
Record Dates: First submitted 2022-05-05; First posted 2022-06-02 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2023-09

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: Probiotic; Non-Alcoholic Fatty Liver Disease; gut microbiota
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Control Groups; Probiotics

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trail
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator): Subjects received two placebo sachets per day
  Interventions: Other: Placebo
- Probiotic group (Experimental): Subjects received two probiotic sachets per day
  Interventions: Dietary Supplement: Probiotics

INTERVENTIONS:
Other: Placebo — Same Additives to Probiotic group but replace probiotics with Corn starch and Maltodextrin.
  Other Names: Control group
  Arms: Placebo group
Dietary Supplement: Probiotics — Multi-strain probiotic supplement includes Lactobacillus reuteri GMNL-263 (heat-killed) and GMNL-89 (alive) and Lactobacillus rhamnosus GMNL-74 ( alive).
  Other Names: Test group
  Arms: Probiotic group

SUMMARY:
In this study, the improvement of the clinical status of early-stage non-alcoholic fatty liver disease (NAFLD) patients after the probiotic intervention will be assessed. And the mechanism of probiotics to prevent the progression of illness would be investigated. The chronic inflammation status, systemic oxidative stress, metabolism of carbohydrates and lipid, and gut microbiota of NAFLD patients will also be analyzed.

DETAILED DESCRIPTION:
Uncontrolled NAFLD evolves in Non-Alcoholic SteatoHepatitis (NASH), cirrhosis and liver cancer. Early intervention to prevent the progression of illness of NAFLD is very important. From 2005 to 2018, 15 clinical trials concluded that multiple-strain probiotics significantly reduced the liver inflammation index and blood lipids in NAFLD patients. Many reports indicated that NAFLD-associated risk factors, such as chronic inflammation, oxidative stress, insulin resistance, dyslipidemia, and obesity are closely correlated with gut microbiota. Some substances (such as endotoxin and alcohol) produced by harmful gut bacteria caused the progression of the illness of NAFLD.

Three strains are Genmont® Normal Lactobacillus (GMNL) which were divided from natural environments, included Lactobacillus reuteri GMNL-263 (heat-killed) and GMNL-89 (alive) and Lactobacillus rhamnosus GMNL-74 ( alive). They are all isolated from the gastrointestinal tract of healthy Taiwanese and were known as common food material worldwide. The previous clinical research on probiotic consumption in type 2 Diabetes mellitus patients under normal drug treatment was conducted in Changhua Christian Hospital. Results showed that L. reuteri GMNL-263 was able to stabilize the weight and blood pressure of patients. L. reuteri GMNL-89 had a stable effect on glycated hemoglobin. There was no adverse reaction when probiotics combining with type 2 diabetes drugs. Meanwhile, L. rhamnosus GMNL-74 was observed to reduce weight gain in obese mice. In this clinical study, The anti-liver inflammation effect of consumption of Lactobacillus sachet in NAFLD patients will be demonstrated at baseline, 3 months and 6 months. In this clinical study, the anti-liver inflammation effect of consumption of Lactobacillus sachet in NAFLD patients will be demonstrated at baseline, 3 months and 6 months to understand the impact of the probiotics on NAFLD. Since the treatment of fatty liver should focus on controlling weight, blood sugar, and blood fat, the relevant clinical indexes will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Nonalcoholic fatty liver disease (NALFD) by ultrasound.
* The range of Alanine aminotransferase (ALT) blood test is 60-300 U/L

Exclusion Criteria:

* Alcoholic consumption (Female ≥ 10g/day or Male ≥ 20g/per)
* Patients with liver diseases, HBV(hepatitis B virus), HCV(hepatitis C virus), Primary Biliary Cholangitis.
* Autoimmune system disease
* Wilson's disease
* Hereditary hemochromatosis
* Patients with uncontrolled malignancy
* The subject had previously received weight reduction surgery
* Taking Antibiotics, probiotics, or any other drugs that affect NAFLD or glucose and lipid metabolism in past 2 months
* Pregnant or lactating female patients
* Patient who have severe allergy to soybeans or peanuts

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Serum ALT (Alanine Aminotransferase) level at baseline | baseline
  The number of patients will be enrolled with the concentration of ALT (Alanine Aminotransferase) ranging from 60 to 300 U/mL in serum.
Change from baseline in Serum ALT (Alanine Aminotransferase) level at 3-months | 3-months
  Fasting blood samples will be collected to examine the variation of ALT (Alanine Aminotransferase).
Change from baseline in Serum ALT (Alanine Aminotransferase) level at 6-months | 6-months
  Fasting blood samples will be collected to examine the variation of ALT (Alanine Aminotransferase).

SECONDARY OUTCOMES:
Change from baseline in BMI (Body Mass index) at 3-months | 3-months
  BMI will be calculated with weight and height combined in kg/m^2, the weight will be measured in kilograms and the height will be recorded in centimeters.
Change from baseline in BMI (Body Mass index) at 6-months | 6-months
  BMI will be calculated with weight and height combined in kg/m^2, the weight will be measured in kilograms and the height will be recorded in centimeters.
Change from baseline in Waist and hip circumference at 3-months | 3-months
  Waist and hip circumference will take down in centimeters.
Change from baseline in Waist and hip circumference at 6-months | 6-months
  Waist and hip circumference will take down in centimeters.
Change from baseline in blood pressure at 3-months | 3-months
  The unit of measurement of blood pressure is mmHg. Both systolic and diastolic blood pressure will be measured.
Change from baseline in blood pressure at 6-months | 6-months
  The unit of measurement of blood pressure is mmHg. Both systolic and diastolic blood pressure will be measured.
Change from baseline in the progress of the non-alcoholic fatty liver disease at 3-months | 3-months
  Utilizing abdominal ultrasound to detect the progress of Non-alcoholic fatty liver disease (NAFLD).
Change from baseline in the progress of the non-alcoholic fatty liver disease at 6-months | 6-months
  Utilizing abdominal ultrasound to detect the progress of Non-alcoholic fatty liver disease (NAFLD).
Change from baseline in levels of AST(Aspartate Aminotransferase) at 3-months | 3-months
  Fasting blood samples will be collected to examine changes from baseline in AST(Aspartate Aminotransferase) in IU/L at 3-months.
Change from baseline in levels of AST(Aspartate Aminotransferase) at 6-months | 6-months
  Fasting blood samples will be collected to examine changes from baseline in AST(Aspartate Aminotransferase) in IU/L at 6-months.
Change from baseline in the level of γ-GT (γ-Glutamyl Transpeptidase) at 3-months | 3-months
  Fasting blood samples will be collected to examine changes from baseline in γ-GT (γ-Glutamyl Transpeptidase) in IU/L at 3-months.
Change from baseline in the level of γ-GT (γ-Glutamyl Transpeptidase) at 6-months | 6-months
  Fasting blood samples will be collected to examine changes from baseline in γ-GT (γ-Glutamyl Transpeptidase) in IU/L at 6-months.
Change from baseline in the level of BUN (Blood Urea Nitrogen) at 3-months | 3-months
  Fasting blood samples will be collected to examine changes in BUN(Blood Urea Nitrogen) from baseline in mg/dL at 3-months.
Change from baseline in the level of BUN (Blood Urea Nitrogen) at 6-months | 6-months
  Fasting blood samples will be collected to examine changes from baseline in BUN(Blood Urea Nitrogen) in mg/dL at 6-months.
Change from baseline in the level of CRE (Creatinine) at 3-months | 3-months
  Fasting blood samples will be collected to examine changes from baseline in CRE(Creatinine) in mg/dL at 3-months.
Change from baseline in the level of CRE (Creatinine) at 6-months | 6-months
  Fasting blood samples will be collected to examine changes from baseline in CRE(Creatinine) in mg/dL at 6-months.
Change from baseline in levels of FBS (Fasting Blood Sugar) at 3-months | 3-months
  Fasting blood samples will be collected to examine changes from baseline in FBS(Fasting Blood Sugar) in mg/dL at 6-months.
Change from baseline in the level of FBS (Fasting Blood Sugar) at 6-months | 6-months
  Fasting blood samples will be collected to examine changes from baseline in FBS(Fasting Blood Sugar) in mg/dL at 6-months.
Change from baseline in levels of HbA1c (Hemoglobin A1C) at 3-months | 3-months
  Fasting blood samples will be collected to investigate the levels of HbA1c(Hemoglobin A1C) in % from baseline at 3-months.
Change from baseline in levels of HbA1c (Hemoglobin A1C) at 6-months | 6-months
  Fasting blood samples will be collected to investigate the levels of HbA1c(Hemoglobin A1C) in % from baseline at 6-months.
Change from baseline in levels of serum insulin at baseline | 3-months
  Fasting blood samples will be collected to examine variation in serum insulin in uIU/mL from baseline at 3-months.
Change from 3-months in levels of serum insulin at baseline | 6-months
  Fasting blood samples will be collected to examine variation in serum insulin in uIU/mL from baseline at 6-months.
Change from Baseline in levels of HOMA-IR (Homeostatic Model Assessment for Insulin Resistance) at 3-months | 3-months
  HOMA-IR(Homeostatic Model Assessment for Insulin Resistance) will be calculated with insulin and glucose. (HOMA-IR=(insulin (mIU/L) and glucose (mg/dl))/405)
Change from baseline in levels of HOMA-IR (Homeostatic Model Assessment for Insulin Resistance) at 6-months | 6-months
  HOMA-IR(Homeostatic Model Assessment for Insulin Resistance) will be calculated with insulin and glucose. (HOMA-IR=(insulin (mIU/L) and glucose (mg/dl))/405)
Change from baseline in levels of TC (Total Cholesterol) at 3-months | 3-months
  Fasting blood samples will be collected to examine variation from baseline in (Total Cholesterol) in mg/dL at 3-months.
Change from baseline in levels of TC (Total Cholesterol) at 6-months | 6-months
  Fasting blood samples will be collected to examine variation from baseline in (Total Cholesterol) in mg/dL from baseline at 6-months.
Change from baseline in level of HDL (High density lipoprotein) at 3-months | 3-months
  Fasting blood samples will be collected to examine variation from baseline in HDL(High density lipoprotein) in mg/dL at 3-months.
Change from baseline in level of HDL (High density lipoprotein) at 6-months | 6-months
  Fasting blood samples will be collected to examine variation from baseline in HDL(High density lipoprotein) in mg/dL at 6-months.
Change from baseline in level of LDL (Low density lipoprotein) at 3-months | 3-months
  Fasting blood samples will be collected to examine variation from baseline in LDL(Low density lipoprotein) in mg/dL at 3-months.
Change from baseline in level of LDL (Low density lipoprotein) at 6-months | 6-months
  Fasting blood samples will be collected to examine variation from baseline in LDL(Low density lipoprotein) in mg/dL at 6-months.
Change from baseline in level of TG (Triglyceride) at 3-months | 3-months
  Fasting blood samples will be collected to examine variation from baseline in TG(Triglyceride) in mg/dL to 3-months.
Change from baseline in level of TG (Triglyceride) at 6-months | 6-months
  Fasting blood samples will be collected to examine variation from baseline in TG(Triglyceride) in mg/dL to 6-months.
Change from baseline in level of hs-CRP (high-sensitivity C-reactive protein) at 3-months | 3-months
  Blood samples will be collected to examine variation from baseline in hs-CRP(high-sensitivity C-reactive protein) in mg/dL at 3-months.
Change from baseline in level of hs-CRP (high-sensitivity C-reactive protein) at 6-months | 6-months
  Blood samples will be collected to examine variation from baseline in hs-CRP(high-sensitivity C-reactive protein) in mg/dL at 6-months.
Change from baseline in level of TNF-α (Tumor necrosis factor-α) at 3-months | 3-months
  Blood samples will be collected to examine variation from baseline in TNF-α (Tumor necrosis factor-α) in pg/mL at 3-months.
Change from baseline in level of TNF-α (Tumor necrosis factor-α) at 6-months | 6-months
  Blood samples will be collected to examine variation from baseline in TNF-α (Tumor necrosis factor-α) in pg/mL at 6-months.
Change from baseline in level of IL-1β (Interleukin-1 β) at 3-months | 3-months
  Blood samples will be collected to examine variation from baseline in IL-1β(Interleukin-1 β) in pg/mL at 3-months.
Change from baseline in level of IL-1β (Interleukin-1 β) at 6-months | 6-months
  Blood samples will be collected to examine variation from baseline in IL-1β(Interleukin-1 β) in pg/mL at 6-months.
Change from baseline in level of IL-6 (Interleukin-6) at 3-months | 3-months
  Blood samples will be collected to examine variation from baseline in IL-6(Interleukin-6) in pg/mL at 3-months.
Change from baseline in level of IL-6 (Interleukin-6) at 6-months | 6-months
  Blood samples will be collected to examine variation from baseline in IL-6(Interleukin-6) in pg/mL at 6-months.
Change from baseline in level of LPS (Lipopolysaccharides) at 3-months | 3-months
  Blood samples will be collected to examine variation from baseline in LPS(Lipopolysaccharides) in mg/dL at 3-months.
Change from baseline in level of LPS (Lipopolysaccharides) at 6-months | 6-months
  Blood samples will be collected to examine variation from baseline in LPS(Lipopolysaccharides) in mg/dL at 6-months.
Change from baseline in level of Leptin at 3-months | 3-months
  Blood samples will be collected to examine variation from baseline in Leptin in pg/mL at 3-months.
Change from baseline in level of Leptin at 6-months | 6-months
  Blood samples will be collected to examine variation from baseline in Leptin in pg/mL at 6-months.
Change from baseline in level of Adiponectin at 3-months | 3-months
  Blood samples will be collected to examine variation from baseline in Adiponectin in pg/mL at 3-months.
Change from baseline in level of Adiponectin at 6-months | 6-months
  Blood samples will be collected to examine variation from baseline in Adiponectin in pg/mL at 6-months.
Change from baseline in the level of SCFA (Short Chain Fatty Acids) at 6-months | 6-months
  Blood samples will be collected to examine variation from baseline in SCFA (Short Chain Fatty Acids) in ug/mL at 6-months.
Change from baseline in the level of TMAO (Trimethylamine N-oxide) at 6-months | 6-months
  Blood samples will be collected to examine variation from baseline in TMAO (Trimethylamine N-oxide) in μmol/L at 6-months.
Change from baseline in Self-questionnaire of Diet and lifestyle assessments at 6-months | 6-months
  The questionnaire will record dietary/drink preferences and other habits by the subject himself /herself, the content of the questionnaire includes vegetarian or not, the frequency if intake of tea, dairy, coffee or yakult intake, smoking habits, betel nuts intake and alcohol consumption.
Change from baseline in self-record of the International physical activity questionary (IPAQ) in physical assessment at 6-months | 6-months
  The questionnaire will be finished to record the laborious activity by the subject himself /herself before and after the treatment.
Change from baseline in gut microbiota at 6-months | 6-months
  The analysis of Gut microbiota will utilize DNA sequencing to investigate the intestinal microbiota through stool samples in subjects with NAFLD at 6-months.

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Yang Chang, PhD, Principal Investigator — Fu Jen Catholic University Hospital
Locations (1):
- Fu Jen Catholic University Hospital, New Taipei City, Taiwan